CLINICAL TRIAL: NCT02871349
Title: Trial of Propranolol in Children and Youth With Autism Spectrum Disorder and Predictors of Response
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Beversdorf, Professor, Department of Radiology & Thompson Center for Autism & Neurodevelopmental Disorders, University of Missouri-Columbia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2005213
Record Dates: First submitted 2016-08-15; First posted 2016-08-18 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Propranolol; Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Propanolol and MRI (Experimental): Participants will receive propranolol via oral capsule, crushed tablet, or liquid daily. The drug dosage will be titrated slowly to ensure the drug is tolerated well. Those aged 15-24 will have an MRI before starting drug.
  Interventions: Drug: Propranolol; Device: Magnetic Resonance Imaging (MRI)
- Placebo and MRI (Placebo Comparator): Participants will receive placebo via oral capsule, crushed tablet, or liquid daily. Those aged 15-24 will have an MRI before starting drug.
  Interventions: Drug: Placebo; Device: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Drug: Propranolol — Propanolol will be given on a titration schedule in which participants will begin with small doses (single capsules) of the drug and increase to a larger dosage (divided over 3 capsules) over the course of three weeks. Participants aged 15-24 years will undergo an MRI.
  Other Names: Inderal; Hemangeol; Innopran
  Arms: Propanolol and MRI
Drug: Placebo — Placebo will be given in the form preferred by the participant and on the same schedule as the propanolol regime. Participants aged 15-24 years will undergo an MRI.
  Arms: Placebo and MRI
Device: Magnetic Resonance Imaging (MRI) — An MRI will be performed on participants aged 15-24 years.

SUMMARY:
The purpose of this study is to find out how the brain of people with autism is affected by Propranolol. Propranolol is not FDA approved for the treatment of autism. Propranolol is FDA approved for the treatment of heart conditions such as blood pressure

This research is being done because there are currently no drug treatment options for language impairments and social difficulties often experienced by people with autism.

DETAILED DESCRIPTION:
The specific aim of this study is to examine the effects of serial doses of propranolol on social interaction, and secondarily on language tasks, anxiety, adaptive behaviors, and global function in high functioning adults and adolescents with autism in a double-blinded, placebo-controlled trial. The investigators will also examine whether response to treatment can be predicted based upon markers of autonomic functioning, such as skin conductance, heart rate variability (HRV), and the pupillary light reflex (PLR), and whether anxiety can predict treatment response. The hypothesis is that social functioning and language abilities will benefit from serial doses of propranolol, and that those with the greatest degree of autonomic dysregulation, or the lowest functional connectivity, will demonstrate the greatest benefit from the drug.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder diagnosis
* intelligence quotient (IQ) >= 85 (if aged 15-24), >= 75 (if aged 7-14)
* Native English speaker
* Parent or caregiver must older than 18 years and be a native English speaker

Exclusion Criteria:

* Taking Alpha 2 agonists
* Non-autism learning disorder
* Other major psychiatric disorders
* Other neurological disorders
* Major head trauma
* Reaction to adhesives
* Diabetes
* Reactive airway disease
* Thyroid disease
* Bradyarrhythmias
* Unexplained syncope
* Pregnancy
* Possible interacting drugs
* Underweight (<20kg if aged 7-14 years)
* Factors affecting ability to have an MRI (if aged 15-24 years)

Ages: 7 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 69 (Actual)
Dates: Start 2016-08; Primary Completion 2020-08 (Actual); Study Completion 2020-08 (Actual)

PRIMARY OUTCOMES:
Change in General Social Outcomes Measure (GSOM) Assessment | Day 1, 6 weeks, 12 weeks

SECONDARY OUTCOMES:
Change in Social Responsiveness Scale (SRS-2) | Day 1, 6 weeks, 12 weeks
Change in score on Anagrams test | Day 1, 6 weeks, 12 weeks
  For those aged 15-24 only
Change in Semantic fluency test results | Day 1, 6 weeks, 12 weeks
  For those aged 15-24 only
Change Clinical Global Impression surveys | Day 1, 6 weeks, 12 weeks
Change in Autism Impact Measure (AIM) | Day 1, 6 weeks, 12 weeks
Change in Clinical Evaluation of Language Fundamentals (CELF-5) assessment | Day 1, 6 weeks, 12 weeks
Change in Vineland Adaptive Behavior Scales (VABS-2) assessment | Day 1, 6 weeks, 12 weeks
Change in score on Aberrant Behavior Checklist (ABC) | Day 1, 6 weeks, 12 weeks
Change in gastrointestinal symptomology | Day 1, 1 week, 2 weeks, 6 weeks, 12 weeks
  Rome IV Diagnostic Questionnaire on Pediatric Functional Gastrointestinal Disorders (R4PDQ-child) and Rome IV Diagnostic Questionnaire (R4DQA) for adults

OTHER OUTCOMES:
Change in Companion Animal Bonding Scale | Day 1, 6 weeks, 12 weeks
Change in Sympathetic Tone & Anxiety Measurements | Day 1, 12 weeks
  Pupillary light reflex, heart rate, heart rate variability, skin conductance, and blood pressure
Changes in salivary cortisol | Day 1, 6 weeks, 12 weeks
Changes in Sensory Over-Responsivity questionnaire | Day 1, 6 weeks, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: David Q Beversdorf, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- Thompson Center for Autism & Neurodevelopmental Disorders, Columbia, Missouri, United States

DOCUMENTS (1):
  • Study Protocol (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT02871349/Prot_000.pdf